CLINICAL TRIAL: NCT03109951
Title: Abnormal Blood Sugar Tests in Diabetic Patients During Colonoscopy Preparation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic Kwandong University (Other)
Responsible Party: Principal Investigator, Myong Ki Baeg, Assistant professor, Catholic Kwandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IS16OASI0026
Record Dates: First submitted 2017-04-03; First posted 2017-04-12 (Actual); Results first posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Type 2 Diabetes Mellitus; Colonoscopy
Keywords: Type 2 diabetes; colonoscopy; hypoglycemia; hyperglycemia; polyethylene glycol
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia; Hyperglycemia

STUDY DESIGN:
Intervention Model Description: Single group
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diabetes group (Other): Type 2 diabetes patients undergoing colonoscopy with preparation with 2L of polyethylene glycol.
  Interventions: Drug: Colonoscopy preparation using polyethylene glycol

INTERVENTIONS:
Drug: Colonoscopy preparation using polyethylene glycol — Colonoscopy preparation using standard preparation with 2L of polyethylene glycol.
  Other Names: Have not taken diabetes medication since 6pm of the day before colonoscopy.; Have fasted since 6pm of the day before colonoscopy.

SUMMARY:
Type 2 diabetes is rapidly increasing globally and has been associated with an increased risk of colorectal cancer. Therefore, the numbers of diabetic patients who will undergo colonoscopic screening are expected to grow exponentially. Colonoscopic preparation entails prolonged fasting, cessation of anti-diabetic medication and ingestion of preparation medications. This may put the diabetic patient at risk of potentially dangerous hypo- or hyperglycemia. However, studies regarding the safety of colonoscopic preparation in diabetic are lacking. In this study, the investigators aim to discover the prevalence of abnormal glucose levels in diabetic patients who undergo colonoscopy. The investigators also aim to find out risk factors for abnormal glucose levels and develop a safe preparation protocol.

DETAILED DESCRIPTION:
1. Type 2 diabetes subjects who will undergo colonoscopy will be prospectively enrolled when visiting the outpatient clinic.
2. Subjects will be instructed to fast from 6pm of the day before colonoscopy.
3. Subjects will be instructed to abstain from diabetes medication while the subjects fast.
4. Subjects who are scheduled to undergo colonoscopy in the morning will take colonoscopy preparation medication (2L (liter) of polyethylene glycol with ascorbic acid) in a split dose (i.e. 1L from 8-10 pm of the day before colonoscopy and 1L 4-6 hours before colonoscopy). Those who will undergo colonoscopy in the afternoon will take 2L of the preparation medication 6 hours before colonoscopy.
5. Subjects will be instructed to take the preparation medication at rate of 250 mL every 10 to 15 minutes.
6. Upon arrival at the endoscopy center of International St. Mary's hospital, subjects will be given a self-administered questionnaire which will ask about their age, gender, duration of diabetes, type of diabetes medication, time of last diabetes medication taken, knowledge of hypo/hyperglycemia symptoms, previous hypo/hyperglycemia experience, self-treatment of hypoglycemia (if done), total amount of colonoscopy preparation medication ingested, total fasting time and time of last preparation medication ingested.
7. Subjects will have vital signs (blood pressure, heart rate) taken and their capillary glucose levels checked using the Accu-Chek Performa.
8. Any subjects with capillary glucose levels <70mg/dL or >250mg/dL will be reported to the attending physician. Those with an initial glucose level <70mg/dL will be given a piece of candy and have their glucose rechecked in 10 mins. Subjects will be asked if the hypoglycemic symptoms (if any) have abated. Those with a glucose level >250mg/dL will undergo hydration with normal saline at 120 ml/Hr. Those who do not respond to treatment or are in critical condition will be moved to the Emergency department for treatment. Subjects who respond to treatment will have their glucose levels checked after colonoscopy before undergoing discharge. Those with abnormal levels upon follow-up testing will be sent to either the endocrinology outpatient clinic or the emergency room depending on their clinical severity.
9. All data will be recorded by initials with patient identities masked. All data will be kept in a locked and secure location by the principal investigator.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Between ages of 20-75
* Undergo colonoscopy at International St. Mary's Hospital

Exclusion Criteria:

* Type 1 diabetes patients
* Did not undergo colonoscopy preparation
* Did not meet fasting requirements
* Have known current infectious diseases
* Have known cancer and/or are under cancer treatment
* Are under intravenous fluid therapy during colonoscopy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2017-03-25 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myong Ki Baeg, MD, PhD, Principal Investigator — International St. Mary's Hospital, Catholic Kwandong University
Locations (1):
- International St.Mary's Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vann MA. Perioperative management of ambulatory surgical patients with diabetes mellitus. Curr Opin Anaesthesiol. 2009 Dec;22(6):718-24. doi: 10.1097/ACO.0b013e3283310f51. PMID 19696663
- [Background] Kollarits CR, Kendrick RM, Guess M. Perioperative treatment of patients with diabetes having eye surgery with local anesthesia in an ambulatory facility. Ophthalmic Surg Lasers Imaging. 2004 May-Jun;35(3):185-8. PMID 15185785
- [Background] Joshi GP, Chung F, Vann MA, Ahmad S, Gan TJ, Goulson DT, Merrill DG, Twersky R; Society for Ambulatory Anesthesia. Society for Ambulatory Anesthesia consensus statement on perioperative blood glucose management in diabetic patients undergoing ambulatory surgery. Anesth Analg. 2010 Dec;111(6):1378-87. doi: 10.1213/ANE.0b013e3181f9c288. Epub 2010 Oct 1. PMID 20889933
- [Background] Yao J, Zhang W, Chen J, Zhang G, Zheng S. Enteral nutrition before bowel preparation improves the safety of colonoscopy in the elderly. Turk J Gastroenterol. 2013;24(5):400-5. doi: 10.4318/tjg.2013.0638. PMID 24557963

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: None noted as this was a single-arm study.
Period: Overall Study
Arm/Group | Diabetes Group
Started | 187
Completed | 187
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diabetes Group
Number analyzed (Participants) | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 117
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Korean Ethnicity | 187
Region of Enrollment [Number; unit: participants]
  South Korea | 187
Fasting glucose level [Mean (Standard Deviation); unit: mg/dL] | 135.9 (33.1)
Number of polyps [Mean (Standard Deviation); unit: polyps] | 1.3 (2.0)
Number of adenomas [Mean (Standard Deviation); unit: adenomas] | 1.1 (1.8)
Number of advanced adenomas [Mean (Standard Deviation); unit: advanced adenomas] | 0.2 (0.5)
Diabetes history [Mean (Standard Deviation); unit: years] — Previous Diabetes history before study enrollment.
  years | 7.3 (7.9)
Fasting period [Mean (Standard Deviation); unit: hours] — Time(hours) from last meal intake to colonoscopy start.
  hours | 19.2 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Abnormal Glucose Levels After Colonoscopic Preparation
Description: Count of patients with Serum glucose levels < 70mg/dL or >250mg/dL
Time Frame: 30 minutes before colonoscopy
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetes Group
Number analyzed (Participants) | 187
Participants
  Number of hyperglycemia subjects | 2
  Number of hypoglycemia subjects | 0
  Number of subjects without hypo or hyperglycemia | 185

2. Secondary Outcome: Cognition of Hypoglycemic Symptoms
Description: Subjects awareness of hypoglycemic symptoms - by questionnaire 96 subjects were aware of hypoglycemic symptoms and could recognize them.
Time Frame: 30 minutes before colonoscopy
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetes Group
Number analyzed (Participants) | 187
Participants | 96

3. Secondary Outcome: Number of Participants With Self-treatment and Relief of Hypoglycemic Symptoms
Description: Discover if self-treatment of hypoglycemic symptoms relieves hypoglycemia and associated symptoms
Time Frame: From colonoscopy preparation beginning to day 1 after colonoscopy
Population: 4 subjects reported hypoglycemia symptoms. All recovered through self-treatment (e.g. drinking juice or taking candy).
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetes Group
Number analyzed (Participants) | 187
Participants | 4

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 1 month.
Arm/Group | Diabetes Group
All-Cause Mortality (participants affected / at risk) | 0/187
Serious Adverse Events (participants affected / at risk) | 0/187
Other Adverse Events (participants affected / at risk) | 0/187

LIMITATIONS AND CAVEATS:
Smaller number of subjects than anticipated due to poor enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/51/NCT03109951/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/51/NCT03109951/ICF_001.pdf